CLINICAL TRIAL: NCT01566409
Title: Maintenance Treatment With Polyethylene Glycol 3350 for Children With Constipation. A Randomized, Placebocontrolled Intervention Study
Brief Title: Maintenance Treatment for Children With Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Line Modin (Other)
Collaborators: University of Southern Denmark (Other); Kolding Sygehus (Other)
Responsible Party: Sponsor-Investigator, Line Modin, Medical doctor, Vejle Hospital
Organization: Vejle Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MainCon
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Results first posted 2016-09-28 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-08

CONDITIONS: Constipation
Keywords: Constipation; Maintenance treatment; Ultrasound of rectum
MeSH Terms: conditions — Constipation | interventions — polyethylene glycol 3350

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active maintenance treatment (Active Comparator)
  Interventions: Drug: Polyethylene glycol 3350
- Placebo maintenance treatment (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Polyethylene glycol 3350 — Powder for solution. Each sachet contains 13.125 g of macrogol 3350. Disimpaction dosage consists of 1,5 g/kg, maintenance treatment are adjusted according til the Bristol stool chart. The drug can be taken at anytime of the day and can also be divided. Treatment duration up to ½ year.
  Other Names: Movicol; Movicol junior; Moxalole; Lacrofarm
  Arms: Active maintenance treatment
Other: Placebo — Placebo will be manufactured and packaged as a powder to make it identical to the bags with the PEG 3350. The powder will comprise of a non-active substance, like a mild rehydration solution, which is a composition consisting of salt and sugar.
  Arms: Placebo maintenance treatment

SUMMARY:
Constipation is a common problem among children. The majority of children suffering from constipation have no underlying disease. Although constipation has no basis in underlying disease, it often leads to a reduced quality of life of children who are on par with or worse than for children suffering from serious diseases such as cardiovascular and rheumatic diseases.

Despite the high frequency of constipation among children, little is known about the causes and treatment of constipation.

Treatment consists of symptomatic treatment with various laxatives. Movicol and Movicol junior has proven very effective and are therefore widely used in children as disimpaction and maintenance treatment. There is currently no research to prove the need for and length of maintenance treatment with laxative medications in children.

The purpose is to examining the effectiveness of maintenance treatment with Movicol. Additional til study will examine how the anal diameter change during a course of treatment and the degree to which it can be used as an indicator of treatment efficacy.

The study will test the following:

• What is the effect of maintenance treatment with PEG compared to placebo?

The results from this study are expected to form the basis for an evidence-based approach to the use of maintenance therapy and the use of ultrasound of the rectum in children with constipation.

ELIGIBILITY:
Inclusion Criteria:

* Children between 2 and 16 years and referral to our out patient clinic with either constipation or fecal incontinence.
* Patients must fulfill the Rome III criteria of constipation, which mean they must have at least 2 of the following characteristics: fewer than 3 bowel movements weekly, more than 1 episode of fecal incontinence weekly, large stools in the rectum by digital rectal examination or palpable on abdominal examination, occasional passing of large stools, display of retentive posturing and withholding behavior, and painful defecation.

Exclusion Criteria:

* Children with known organic causes of constipation, including Hirsprung disease, spinal and anal congenital abnormalities, previous surgery on the colon, inflammatory bowel disease, allergy and metabolic or endocrine diseases.
* Children receiving drugs known to affect bowel function during a 2 month period before initiation.
* The healthy control group consists of children with no history of constipation (Rome III), urinary incontinence, urinary tract infections, fecal incontinence, laxative use or any other disease affecting the digestive system.
* Children receiving medications known to affect bowel function are excluded from the study.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 115 (Actual)
Dates: Start 2013-09; Primary Completion 2015-04 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Line Modin, Kolding, Denmark

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Maintenance Treatment | Placebo Maintenance Treatment
Started | 49 | 53
Completed | 47 | 48
Not Completed | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Maintenance Treatment | Placebo Maintenance Treatment | Total
Number analyzed (Participants) | 49 | 53 | 102
Age, Customized [Median (Full Range); unit: years] | 6.2 [2.5 to 12.3] | 6.1 [2.0 to 15.1] | 6.1 [2.0 to 15.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 27 | 45
  Male | 31 | 26 | 57
Region of Enrollment [Number; unit: participants]
  Denmark | 49 | 53 | 102

OUTCOME MEASURES:

1. Primary Outcome: Treatment Recovery
Description: Recovery is defined as the child having no symptoms of constipation according to the Rome III criteria.
Time Frame: ½ year
Measure: Number; unit: participants
Arm/Group | Active Maintenance Treatment | Placebo Maintenance Treatment
Number analyzed (Participants) | 49 | 53
participants | 33 | 19
Statistical Analysis 1: Comparison: Active Maintenance Treatment vs Placebo Maintenance Treatment; Test type: Non-Inferiority or Equivalence — The required sample size was based on a projected treatment success in the PEG group of 60%. With a power in excess of 80% and a critical level of significance of 0.05, 45 children were needed in each group to detect a 50% reduction in treatment effect in the placebo group, corresponding to 30% recovers without active maintenance treatment. Because of an expected drop-out rate of 25%, we aimed at including 115 children; p = 0.024, Regression, Logistic

2. Secondary Outcome: Usage of Laxative
Time Frame: ½ year
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Active Maintenance Treatment | Placebo Maintenance Treatment
Serious Adverse Events (participants affected / at risk) | 1/49 | 0/53
Other Adverse Events (participants affected / at risk) | 25/49 | 32/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Maintenance Treatment (N=49) | Placebo Maintenance Treatment (N=53)
Broken arm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Maintenance Treatment (N=49) | Placebo Maintenance Treatment (N=53)
abdominal pain (Gastrointestinal disorders) | 6 (12) | 22 (40)
Bloating (Gastrointestinal disorders) | 1 (12) | 0 (0)
Fever, upper respiratory infektion (Infections and infestations) | 17 (34) | 9 (22)
Headach (Nervous system disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less